CLINICAL TRIAL: NCT02660918
Title: Decreasing Postoperative Pain Following Endometrial Ablation: A Randomized Controlled Trial
Brief Title: Decreasing Postoperative Pain Following Endometrial Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Jordan Klebanoff, Principal Investigator, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35179
Record Dates: First submitted 2016-01-19; First posted 2016-01-21 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Women undergoing endometrial ablation that meet the eligibility criterial will receive a standardized paracervical injection of Bupivacaine 20 mL 0.25% at the completion of the procedure.
  Interventions: Drug: Bupivacaine
- Control (Placebo Comparator): Women undergoing endometrial ablation that meet the eligibility criterial will receive an equal volume standardized paracervical injection of Normal Saline at the completion of the procedure.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Bupivacaine — Paracervical injection of 20 mL 0.25% Bupivacaine at the completion of the procedure
  Other Names: Marcaine, Sensorcaine
  Arms: Treatment
Other: Normal Saline — Equal volume injection of normal saline with the same paracervical technique
  Arms: Control

SUMMARY:
To determine whether paracervical injection of long acting local anesthesia decreases postoperative pain following endometrial ablation under general anesthesia.

DETAILED DESCRIPTION:
Destruction of the endometrial lining to control bothersome uterine bleeding has been implemented since 1937. Currently there are various different 'second generation' energy sources to avert such bleeding, five of which are now approved in the United States. These 5 second generation devices include: Thermachoice/Cavaterm, which use high temperature fluid within a balloon; Microsulis, which applies microwaves; Novasure, which uses bipolar energy; Hydrothermablator, which uses free fluid at high temperatures; ELITT, which uses laser thermotherapy; and HerOption, which uses cryoablation. Patient selection for endometrial ablation is crucial, as it is intended for premenopausal women with normal uterine cavities and no desire for future fertility that are affected by heavy menstrual bleeding. Since the introduction of the initial 'second generation' device in 1997 these modalities have overtaken the industry mostly due to their ease of use and shorter operative times. Regardless, a Cochrane review finds insufficient evidence to prove superiority of these newer modalities over the traditional 'gold standard' resectoscopic technique.

Endometrial ablation has been demonstrated in a variety of settings including outpatient surgical centers as well as physician's offices. Evidence suggests that microwave endometrial ablation under local anesthesia is a safe and acceptable practice. Very often, when endometrial ablation is performed as an outpatient procedure, patients are pre-medicated and then receive a paracervical injection of local anesthesia to control pain intraoperatively. When endometrial ablations are performed as an outpatient procedure through a surgical center, a variety of anesthesia techniques are employed depending on the infrastructure and human and institutional resources available. These techniques may vary from conscious sedation to general anesthesia, all of which have been proven to be acceptable methods.

In this center endometrial ablations are performed as an outpatient procedure under general anesthesia with a variety of induction techniques and intraoperative pain management practices. According to physician preference, patients may receive an additional paracervical injection of local anesthetic before the procedure, immediately after, or not at all. To date, there are no studies evaluating the efficacy of local anesthetic in addition to general anesthesia for patients receiving endometrial ablation to guide physician practice. The purpose of this study is to evaluate the efficacy of local anesthetic, in addition to general anesthesia, in our large, community-based patient population, in meaningfully decreasing postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* English as primary language
* undergoing outpatient endometrial ablation at the Christiana Hospital Surgical Center
* Indication of menorrhagia
* Inication of abnormal uterine bleeding
* Indication of thickened endometrium.

Exclusion Criteria:

* Known malignancy
* weight less than 50 Kg
* amide allergy
* history of chronic pain
* cardiac arrhythmia
* dilaudid/codeine allergy
* history of opioid use
* inability to take opioids by mouth
* uterine anomaly
* previous endometrial ablation
* primary language other than English.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Klebanoff, MD, Principal Investigator — Christiana Hospital
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fergusson RJ, Lethaby A, Shepperd S, Farquhar C. Endometrial resection and ablation versus hysterectomy for heavy menstrual bleeding. Cochrane Database Syst Rev. 2013 Nov 29;(11):CD000329. doi: 10.1002/14651858.CD000329.pub2. PMID 24288154
- [Background] Glasser MH, Heinlein PK, Hung YY. Office endometrial ablation with local anesthesia using the HydroThermAblator system: Comparison of outcomes in patients with submucous myomas with those with normal cavities in 246 cases performed over 5(1/2) years. J Minim Invasive Gynecol. 2009 Nov-Dec;16(6):700-7. doi: 10.1016/j.jmig.2009.06.023. PMID 19896596
- [Background] Wallage S, Cooper KG, Graham WJ, Parkin DE. A randomised trial comparing local versus general anaesthesia for microwave endometrial ablation. BJOG. 2003 Sep;110(9):799-807. PMID 14511961

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 42 | 42
Completed | 41 (Age ineligible) | 41 (Age ineligible)
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control: Women undergoing endometrial ablation that meet the eligibility criteria will receive an equal volume standardized paracervical injection of Normal Saline at the completion of the procedure.
  Normal Saline: Equal volume injection of normal saline with the same paracervical technique
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.29 (5.09) | 43.66 (4.54) | 43.47 (4.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 41 | 39 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 14 | 20
  White | 34 | 25 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Insurance [Count of Participants; unit: Participants]
  None | 0 | 0 | 0
  Medicaid | 4 | 5 | 9
  Medicaire | 1 | 1 | 2
  Other Private | 36 | 35 | 71
Indication for Surgery [Count of Participants; unit: Participants]
  Menorrhagia | 28 | 33 | 61
  Abnormal Uterine Bleeding | 12 | 7 | 19
  Thickened Endometrium | 1 | 0 | 1
  Unknown | 0 | 1 | 1
Radiofrequency ablation [Count of Participants; unit: Participants] | 35 | 33 | 68
Hydrothermoablation [Count of Participants; unit: Participants] | 2 | 7 | 9
Thermachoice balloon [Count of Participants; unit: Participants] | 0 | 0 | 0
Minerva Abltion [Count of Participants; unit: Participants] | 1 | 1 | 2
Previous ceasrean delivery [Count of Participants; unit: Participants] | 12 | 13 | 25
Previous tubal ligation [Count of Participants; unit: Participants] | 10 | 13 | 23
Previous myomectomy [Count of Participants; unit: Participants] | 1 | 1 | 2
Previous dilation and curettage [Count of Participants; unit: Participants] | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Score
Description: Pain will be assessed using a 10 point visual analog scale. On the scale 0 represented no pain and 10 represented the highest pain level. Eligibility for analgesia was available for patients who reported pain higher than 5 out of 10 on the scale.
  Pain levels were assessed by trained nursing staff blinded to the study. Lower numbers on the 10 point scale represented a positive outcome.
  Patients
Time Frame: Immediate postoperatively through 8 hours post operation.
Population: not avaialble
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 41 | 41
units on a scale
  1 Hour Postoperative Pain Score | 2.71 (2.47) | 1.44 (2.32)
  4 Hours Postoperative Pain Score: number analyzed (Participants) | 38 | 37
  4 Hours Postoperative Pain Score | 3.37 (2.48) | 2.81 (2.22)
  8 Hours Postopeartive Pain Score: number analyzed (Participants) | 38 | 37
  8 Hours Postopeartive Pain Score | 2.47 (2.17) | 2.24 (1.83)

2. Primary Outcome: Intraoperative Total Blood Loss
Description: Amount of operative blood lost measured in milliliters
Time Frame: Intraoperative
Population: Data was only available for 37 patients in the Control group and 33 patients in the Treatment group
Measure: Median (Standard Deviation); unit: cc
Arm/Group | Control | Treatment
Number analyzed (Participants) | 37 | 33
cc | 6.38 (3.7) | 7.15 (6.06)

3. Primary Outcome: Remaining Tylenol Tablets With Codeine Not Taken at the End of Day 1 Following Discharge
Description: All patients were given 10 tablets of Tylenol with codeine upon discharge for pain. This Outcome measure details the remaining number of tablets after day 1.
Time Frame: Postoperative
Population: Data was only available for 38 patients in the Control group and 38 patients in the Treatment group
Measure: Mean (Standard Deviation); unit: Pills
Arm/Group | Control | Treatment
Number analyzed (Participants) | 38 | 38
Pills | 9.18 (.98) | 8.74 (1.52)

4. Secondary Outcome: Occurrence of Intraoperative Complication
Description: This represents any unanticipated complication related to the endometrial ablation.
Time Frame: During Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 41 | 41
Participants
  Bleeding | 0 | 0
  Uterine Perfortaion | 0 | 0
  Failed Ablation | 2 | 1
  Incomplete Ablation | 0 | 0
  Fluid Overload | 0 | 0

5. Secondary Outcome: Postoperative Complication
Description: Any unanticipated complication related to the endometrial ablation.
Time Frame: 1 Day Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 41 | 41
Participants
  Bleeding | 0 | 0
  Infection | 1 | 2
  Hospital Readmission | 0 | 0

6. Secondary Outcome: Postoperative Opioid Administered Following the Procedure But Prior to Discharge.
Description: Narcotic medications administered in the recovery area before the patient was discharged from the Surgicenter.
Time Frame: Predischarge from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 41 | 41
Participants
  Percocet | 3 | 1
  Vicodin | 0 | 0
  Dialudid | 8 | 6
  Roxicodone | 15 | 9
  tylenol with Codeine | 0 | 0

7. Secondary Outcome: Postoperative Toradol
Description: Data was collected on whether or not the patient received Toradol following the endometrial ablation. Toradol is a non-narcotic pain medication.
Time Frame: Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 41 | 41
Participants | 36 | 32

8. Secondary Outcome: Postoperative Anti-emetic
Description: Data was collected on any nausea medicine administered following the endometrial ablation.
Time Frame: Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 41 | 41
Participants
  Benadryl | 2 | 1
  Zofran | 6 | 1
  Reglan | 0 | 0
  Phenergan | 1 | 0

9. Secondary Outcome: Time Between Recovery Initiation and Discharge
Description: Time between arrival to the recovery room after surgery and discharge to home
Time Frame: hours between recovery initiation and discharge
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Control | Treatment
Number analyzed (Participants) | 41 | 41
hours | 1.63 (.73) | 1.59 (.55)

ADVERSE EVENTS:
Time Frame: From recovery through post operative Day 1
Description: Postoperative Infection
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 1/41 | 2/41
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=41) | Treatment (N=41)
Potsoperative Infection (Infections and infestations) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT02660918/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT02660918/ICF_001.pdf